CLINICAL TRIAL: NCT02009137
Title: A Randomized-Controlled Clinical Trial to Evaluate the Efficacy and Safety of Breast Augmentation With EVERA(Korean External Soft Tissue Expansion System) as Compared to AESTES (American External Soft Tissue Expansion
Brief Title: Efficacy and Safety Study of EVERA to Augment Small Breast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chan-Yeong Heo, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E1307-210-002; 06-2013-175-GNSD (Other Grant/Funding Number: GNSD Co.,Ltd)
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Atrophy of Breast
Keywords: small breast; augmentation; breast volume; External Soft Tissue Expansion System(ESTES)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVERA (Experimental): EVERA- korean ESTES system, apply for 12 weeks
  Interventions: Device: EVERA
- ESTES (Active Comparator): ESTES apply for 12 weeks
  Interventions: Device: ESTES

INTERVENTIONS:
Device: EVERA — EVERA apply for 12 weeks
  Arms: EVERA
Device: ESTES — ESTES apply for 12 weeks
  Arms: ESTES

SUMMARY:
Expected Total Number of Subjects

* Level of significance, alfa 0.05
* Power 0.80
* Mean difference between two treatments is assumed 35
* Standard Deviation is assumed 35.
* Follow-up loss is assumed 20%
* N=34(each group:17)

DETAILED DESCRIPTION:
Study design

* single center, randomized, unblind clinical study Medical device
* Investigational Medical Device: EVERA
* Comparator: ESTES Process
* For eligible subjects, investigator apply Standard Deviation or Comparator on the breast
* The Investigational Medical Device is determined by randomization.
* Subjects will be applied for 12 weeks.
* Subjects will receive Patient Compliance Diary
* Subjects will visit the hospital to measure breast volume with VIVID 9i every 2 weeks for 16weeks

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 24 and 40
* BMI of over 20
* Subjects who want to augment breasts
* Subjects who understand the study contents and signed the informed consent
* Subjects who can follow study procedure

Exclusion Criteria:

* Pregnant or Lactating subjects

Ages: 24 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The change in breast volume of the test group and control group | Baseline and 12weeks and 16weeks

SECONDARY OUTCOMES:
Changes in satisfaction level on their breast | Baseline and 12weeks and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chanyeong - Heo, Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National Univ. Bundang Hospital, Seongnam-si, Gumi-dong, Bundang-gu/Gyeonggi-do, South Korea